CLINICAL TRIAL: NCT02722902
Title: Impact of L-Carnitine Infusion on Lipid Induced Insulin Resistance
Brief Title: Carnitine Infusion and Insulin Resistance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No effect of carnitine on lipid induced insulin resistance after n=8 (p=1.00)
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NL56319.068.16
Record Dates: First submitted 2016-02-26; First posted 2016-03-30 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2017-07

CONDITIONS: Glucose Intolerance
Keywords: Metabolic flexibility; Insulin sensitivity
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — Carnitine; soybean oil, phospholipid emulsion; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LIPID + Carnitor (Experimental): intravenous Lipid infusion (IntraLipid) combined with carnitor (L-carnitine) infusion
  L-Carnitine will be administrated intravenously as continuous infusion during the 6-hour hyperinsulinemic euglycemic clamp. The administration will start with a bolus of 15mg/kg for 10 minutes. Subsequently, continuous L-carnitine infusion of 10mg/kg will start for the remaining 350 minutes.
  Intralipid will be administrated intravenously as continuous infusion during the 6-hour hyperinsulinemic euglycemic clamp. The maximum dosage will not exceed 90 mL/h.
  Interventions: Drug: Carnitor; Dietary Supplement: IntraLipid
- LIPID + PLAC (Placebo Comparator): Intravenous Lipid infusion (IntraLipid) combined with placebo infusion (saline)
  Intralipid will be administrated intravenously as continuous infusion during the 6-hour hyperinsulinemic euglycemic clamp. The maximum dosage will not exceed 90 mL/h.
  Interventions: Dietary Supplement: IntraLipid; Dietary Supplement: Placebo
- PLAC (Placebo Comparator): Infusion of saline (no IntraLipid and no carnitor)
  Saline will be administrated intravenously as continuous infusion during the 6-hour hyperinsulinemic euglycemic clamp. The maximum dosage will not exceed 90 ml/h.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Carnitor — CARNITOR® (levocarnitine) is a carrier molecule in the transport of long-chain fatty acids L-Carnitine will be administrated intravenously as continuous infusion during the 6-hour hyperinsulinemic euglycemic clamp. The administration will start with a bolus of 15mg/kg for 10 minutes. Subsequently, continuous L-carnitine infusion of 10mg/kg will start for the remaining 350 minutes.
  across the inner mitochondrial membrane.
  Other Names: L-Carnitine or Levocarnitine
  Arms: LIPID + Carnitor
Dietary Supplement: IntraLipid — Lipid emulsion for infusion
  Arms: LIPID + Carnitor; LIPID + PLAC
Dietary Supplement: Placebo — Saline will be used as placebo
  Other Names: saline
  Arms: LIPID + PLAC; PLAC

SUMMARY:
Insulin resistant subjects and type 2 diabetic patients are characterized by a decreased metabolic flexibility: a reduced capability to switch from fat oxidation in the basal state to carbohydrate oxidation in the insulin-stimulated state. This metabolic inflexibility is an early hallmark in the development of diabetes. Recent evidence suggests that a low carnitine availability may limit acetylcarnitine formation, thereby reducing metabolic flexibility. Thus, when substrate flux in the muscle is high, acetyl-CoA concentrations increase, leading to inhibition of pyruvate dehydrogenase (PDH) and thereby reducing glucose oxidation. The conversion of acetyl-CoA to acetylcarnitine relieves this acetyl-CoA pressure on PDH. To provide more direct insight into the effect of carnitine in preventing metabolic inflexibility and insulin resistance and to further explore the mechanism of action is the focus of this research. Here, we hypothesize that the capacity to form acetylcarnitine may rescue lipid-induced insulin resistance. To this end, insulin resistance will be induced by lipid infusion in healthy volunteers and it will be tested whether carnitine co-infusion can alleviate insulin resistance.

DETAILED DESCRIPTION:
Rationale: Insulin resistant subjects and type 2 diabetic patients are characterized by a decreased metabolic flexibility: a reduced capability to switch from fat oxidation in the basal state to carbohydrate oxidation in the insulin-stimulated state. This metabolic inflexibility is an early hallmark in the development of diabetes. Recent evidence suggests that a low carnitine availability may limit acetylcarnitine formation, thereby reducing metabolic flexibility. Thus, when substrate flux in the muscle is high, acetyl-CoA concentrations increase, leading to inhibition of pyruvate dehydrogenase (PDH) and thereby reducing glucose oxidation. The conversion of acetyl-CoA to acetylcarnitine relieves this acetyl-CoA pressure on PDH. To provide more direct insight into the effect of carnitine in preventing metabolic inflexibility and insulin resistance and to further explore the mechanism of action is the focus of this research. Here, we hypothesize that the capacity to form acetylcarnitine may rescue lipid-induced insulin resistance. To this end, insulin resistance will be induced by lipid infusion in healthy volunteers and it will be tested whether carnitine co-infusion can alleviate insulin resistance.

Objective: The primary objectives are to investigate whether L-carnitine infusion may rescue lipid-induced insulin resistance and whether L-carnitine infusion is improving metabolic flexibility in the state of lipid-induced insulin resistance. Furthermore, a secondary objective is to examine the molecular pathways of carnitine and acetylcarnitine, responsible for muscle insulin sensitivity.

Study design: The current study is an interventional randomized crossover trial in which each subject serves as it owns control. Subjects will be blinded for the intervention.

Study population: n=10, healthy young (18-40 years) male subjects will be included.

Intervention (if applicable): Ten healthy subject will be subjected to the intervention of L-carnitine infusion. To investigate whether L-Carnitine infusion may rescue lipid induced insulin resistance and improve metabolic flexibility three intervention trials are included. The first trial includes lipid infusion combined with L-Carnitine infusion (=LIPID + CAR). In the second trial, L-carnitine infusion will be replaced by placebo infusion in the form of saline (= LIPID + PLAC) in order to investigate the effect of L-Carnitine. During the third trial, lipid infusion will be replaced by infusion of saline and will serve as a control for the lipid infusion (=SALINE + PLAC) and is necessary to investigate to what extend L-carnitine can rescue lipid induced insulin resistance. All three trials will be separated by at least one week. Subjects will be blinded, so no information about the infused substances will be provided to them. The three different trials will be allocated in a random order.

Main study parameters/endpoints: The primary study endpoint is whole body insulin sensitivity, measured by the hyperinsulinemic-euglycemic clamp. Secondary endpoints are maximal acetylcarnitine concentrations after exercise, metabolic compounds in the blood and measurements regarding skeletal muscle metabolism in skeletal muscle tissue obtained by needle biopsies.

ELIGIBILITY:
Inclusion Criteria:

* • Caucasian

  * Healthy (as determined by responsible physician based on a medical questionnaire)
  * Male
  * Age: 18-40 years
  * Normal BMI: 18-25 kg/m2
  * Stable dietary habits
  * No use of medication interfering with investigated study parameters (as determined by responsible physician)

Exclusion Criteria:

* • Female

  * Haemoglobin levels < 7.8 mmol/L
  * Uncontrolled hypertension
  * Use of anticoagulants
  * Engagement in exercise > 3 hours a week
  * Being vegetarian or vegan (because of altered whole body carnitine status)
  * Smoking
  * Alcohol and/or drug abuse
  * Unstable body weight (weight gain or loss > 5kg in the last 3 months)
  * Significant food allergies/intolerances (seriously hampering study meals)
  * Participation in another biomedical study within 1 month before the first study visit, which would possibly hamper our study results
  * Medication use known to hamper subject's safety during the study procedures
  * Medication use known to interfere with investigated study parameters
  * Subjects with contra-indications for MRI
  * Subjects who intend to donate blood during the intervention or subjects who have donated blood less than three months before the start of the study
  * Subjects who do not want to be informed about unexpected medical findings
  * Subjects who do not want that their treating physician is informed

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Whole body insulin sensitivity | 6 hours
  measured as GIR in µmol/kg/min during the stable period of the insulin phase of the clamp.
  * Peripheral insulin sensitivity measured as Rd in µmol/kg/min
Metabolic flexibility | 6-hours
  Change in RER comparing basal and insulin stimulated state during the clamp

SECONDARY OUTCOMES:
Maximal acetylcarnitine concentrations after exercise | 45 minutes
  Measured using 1H-MRS after 30 minutes of cycling at 70% Wmax
glucose concentration in the blood before and during insulin stimulation | 6 hours
  glucose concentration in the plasma will be measured via a blood draw
Carnitine acyltransferase (CRaT) enzyme activity (physiological parameter) | 6 hours
  CRaT activity will be measured in obtained muscle biopsies from the vastus Lateralis muscle using enzyme Activity Assays.
  Measurements will be obtained using 10 ml of sample incubated in 190 ml reaction buffer (50mM Tris-HCl, 1M EDTA, 0.45mM acetyl-CoA, 0.1mM DTNB; pH = 7.8). CrAT specific activity will be determined by measuring the rate of reduction of DTNB (412 nm) by the free CoA liberated from acetylCoA after adding 5mM L-carnitine and monitoring for 10 min
Acylcarnitine profile in the muscle (physiological parameter) | 6 hours
  In muscle tissue obtained via biopsies. Acylcarnitine measurements will be performed using flow injection tandem mass spectrometry
Lipid levels (physiological parameter) | 6 hours
  In muscle tissue obtained via biopsies
free fatty acid in the blood before and during insulin stimulation | 6 hours
  free fatty acid concentration in the plasma will be measured via a blood draw
Triglycerides in the blood before and during insulin stimulation | 6 hours
  Triglycerides wil be measured in the plasma via a blood draw
Insulin in the blood before and during insulin stimulation | 6 hours
  Insulin wil be measured in the plasma via a blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Vera B Schrauwen, Dr, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands